CLINICAL TRIAL: NCT01188395
Title: Bipolar Disorder With Alcoholism in Han Chinese
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Ru-Band Lu/Professor, National Cheng-Kung University Hospital
Other Study IDs: HR-98-002
Record Dates: First submitted 2010-08-23; First posted 2010-08-25 (Estimated); Last update posted 2010-08-25 (Estimated); Status verified 2010-08

CONDITIONS: Bipolar Disorders
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- subtypes of bipolar disorders: Bipolar I Disorder with alcoholism Bipolar I Disorder without alcoholism Bipolar II Disorder with alcoholism Bipolar II Disorder without alcoholism

SUMMARY:
The aim of this study is to explore relation between the comorbidity of different bipolar disorders with alcoholism and neuropsychiatric function and candidate genes. The investigators plan to establish genetic validity for this subtype of alcoholism. In addition, by comparing this subtyped alcoholism to normal control, the investigators plan to examine the genetic validity of such comorbidity. The investigators plan to find specific clinical characteristic from neuropsychiatric aspects of such subtype for future early diagnosis, prediction and prevention.

DETAILED DESCRIPTION:
From family, twin and adoption studies supported a strong hereditary component in unsubtyped alcohol dependency (Cloninger et al., 1981; Reich et al., 1999; Huang et al., 2004). Dopamine, serotonin related genes and ADH, ALDH genes have been considered as candidate genes for alcohol dependency (Goldman, 1995; Reich et al., 1999; Noble et al., 2000). However, both in simple or family-base association studies have generated controversy about the relationship between candidate genes and alcoholism (Edenberg et al., 1998; Reich et al., 1999; Noble et al., 2000). One of the possible explanations may be due to that those studies did not subtype alcohol dependency, even though alcoholism is a complex phenotype with a heterogeneous etiology (Huang et al., 2004; Lu et al., 2005a).

Our previous research results had already categorized AD among Han Chinese in Taiwan into four subtypes, pure alcoholism (Pure ALC), anxiety-depression alcoholism (ANX/DEP ALC), antisocial alcoholism (Antisocial ALC) and mixed type alcoholism (Mixed ALC) （Huang et al., 2004; Lu et al., 2005; Wang et al., 2007）. Except for Mixed ALC, we have established fundamental genetic validity, and confirmed several candidate genes including MAOA、ADH、ALDH、DRD2.

Mixed ALC is categorized by alcoholism comorbid with other psychiatric disorders including schizophrenia and bipolar disorder. Among them all, bipolar disorders most frequently comorbid with alcohol and substance dependence. The high comorbidity between alcohol dependence among patients with bipolar disorder worsens the treatment effect and prognosis. Bipolar disorders are divided into several categories, including bipolar I disorder (BP-I), bipolar II disorder (BP-II), and cyclothymic disorder. Previous literatures have documented that BP-I and BP-II might have different etiology, phenomenology, characteristics and neuropsychiatric functional impairments in the course of the illness (APA, 1994).

The aim of this study is to explore relation between the comorbidity of different bipolar disorders with alcoholism and neuropsychiatric function and candidate genes. We plan to establish genetic validity for this subtype of alcoholism. In addition, by comparing this subtyped alcoholism to normal control, we plan to examine the genetic validity of such comorbidity. We plan to find specific clinical characteristic from neuropsychiatric aspects of such subtype for future early diagnosis, prediction and prevention.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent by patient or legal representative.
2. Male or female patient aged ≧18 and ≦65 years.
3. A diagnosis of Bipolar I or Bipolar II Disorder according to DSM-IV criteria made by a specialist in psychiatry.
4. Patients who were diagnosed with alcohol dependence or abuse according to DSM-IV criteria made by a specialist in psychiatry.

Exclusion Criteria:

1. Patients, except those are Bipolar disorder with alcoholsim who were diagnosed substance abuse/depence
2. Patients with brain injury or regrated neurological diseases
3. Patients who are with I axis major mental illess according to DSM-IV criteria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Bipolar disorders
Sampling Method: Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2009-08; Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Young's Mania Rating Scale (YMRS) | baseline, 3 months
  The severity of manic symptoms of patients will be rated by using YMRS.
Hamilton Depression Rating Scale (HDRS) | baseline, 3 months
  The severity of depressive symptoms of patients will be measured using HDRS.

SECONDARY OUTCOMES:
blood sample | baseline, 3 months
  PCR lab methodology
DNA | baseline
  DRD2 TaqI-A PCR-RFLP ADH2 and ALDH2 PCR-RFLP MAO A genotypes

CONTACTS AND LOCATIONS:
Overall Officials: Ru-Band Lu, MD, Principal Investigator — National Cheng-Kung University Hospital
Locations (1):
- Ru-Band Lu, Tainan, Taiwan